CLINICAL TRIAL: NCT06147791
Title: Risks and Benefits of Using External Scrotal Drainage in Three-piece Penile Prosthesis Implant: a Prospective Randomized Study
Brief Title: Risks and Benefits of Scrotal Drainage in Penile Prosthesis Implant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Mirko Preto, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 833.300
Record Dates: First submitted 2023-10-14; First posted 2023-11-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Group A (drainage) vs Group B (no drainage)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with drainage (Experimental)
  Interventions: Device: External scrotal drainage
- Group without drainage (No Intervention)

INTERVENTIONS:
Device: External scrotal drainage — Application of external scrotal drainage during three-component penile prosthesis placement
  Arms: Group with drainage

SUMMARY:
The goal of this prospective randomized study is to demonstrate if the use of an external scrotal drainage in penile prosthetic surgery can reduce the risk of post-operative complications without increase the risk of infections.

DETAILED DESCRIPTION:
After being informed about the study, all patients give writted informed consent. After that they will be randomized in two groups (A with drainage, B without drainage) using a random sequence generator. Then the patient will undergo the implantation of a three-component penile prosthesis following peri antibiotic prophylaxis with cephalosporins and aminoglycosides, the antibiotic prophylaxis will be continued on the first post-operative day surgery with a cephalosporin. In the group A it will be positioned at the scrotal level (using surgical access or using a second incision) an external drainage (10 Ch in aspiration) for 24 hours. The drainage will be removed on the first post-operative day. The degree of the hematoma will be determined using a 5-point Likert scales already approved in previous cases. Subsequently patients will carry out periodic check-ups at 7, 15 and 30 days after the operation to evaluate the appearance of hematomas and surgical site infection. After that, they will carry out check-ups every month for the first 3 months, then every 3 months for the first year and finally annually up to the fifth year after the intervention. During the clinical check-ups, it will also be defined the time of use of the penile prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed voluntarily according to the rules of good clinical practice (Declaration of Helsinki) and national regulations (Appendix B).
* Genetically male patient.
* Age ≥ 18 years.
* Patient suffering from ED of variable and/or multifactorial etiology.
* Patient suffering from ED not responsive to iPDE-5.
* Patient suffering from unresponsive or non-tolerant ED

Exclusion Criteria:

* Absence of signed written informed consent (Appendix B).
* Age <18 years.
* Genetically female patients.
* Patient with active peno-scrotal infection.
* Patient with active systemic infection.
* Immunosuppressed patient.
* Patient with haematological pathologies that may cause an increased risk of bleeding.
* Patients suffering from Peyronie's Disease who must undergo simultaneous plaque surgery.
* Any condition or situation that, in the opinion of the investigator, places the patient at significant risk, may confound the results of the study, or significantly interfere with the patient's participation in the study.
* The patient declares that it will be impossible for him to participate in follow-up consultations.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative infectious episodes | One month
  Define the number of post-operative infectious episodes in the two study arms.

SECONDARY OUTCOMES:
Post-surgical hematoma | One month
  Define the risk of post-surgical hematoma formation in the two study arms.
Volume of drained material | 24 hour
  Evaluate the volume of drained material in the group with external drainage.
Manipulation of the activation pump | Up to 12 weeks
  Define the time elapsed between surgery and subsequent manipulation of the activation pump in the two study arms, usually 2 weeks.
Activation of the device | Up to 12 weeks
  Define the time elapsed between the surgical intervention and the subsequent activation of the device in the two study arms, usually 3 weeks.
Use of the penile prosthesis | Up to 12 weeks
  Define the time elapsed between surgery and the use of the penile prosthesis for sexual activity in the two study arms, usually 4 weeks after surgery.
Effectiveness of external drainage in subgroups | Up to 12 months
  Compare, through a sub-analysis, the effectiveness of external drainage in different patient populations: heart patients, diabetics, duration of surgery.
  We will test the effectiveness of external drainage in these soubgroups using the IIEF questionnaires.
Effectiveness of external drainage in subgroups | Up to 12 months
  Compare, through a sub-analysis, the effectiveness of external drainage in different patient populations: heart patients, diabetics, duration of surgery.
  We will test the effectiveness of external drainage in these soubgroups using the SSIPI questionnaires.
Effectiveness of external drainage in subgroups | Up to 12 months
  Compare, through a sub-analysis, the effectiveness of external drainage in different patient populations: heart patients, diabetics, duration of surgery.
  We will test the effectiveness of external drainage in these soubgroups using the QoLPSS questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Falcone Mr Marco, Physician, Principal Investigator — Urology
Locations (2):
- Italy (2):
  - SCDU Urologia, Torino, Torino
  - A.O.U. Città della Salute e della Scienza di Torino, Turin, Turin

IPD SHARING:
Plan to Share IPD: No
The data will be shared only among physician participating in the study.